CLINICAL TRIAL: NCT00770848
Title: A Phase 1b/2 Study to Assess the Safety and Efficacy of AMG 102 in Combination With Mitoxantrone and Prednisone in Subjects With Previously Treated Castrate Resistant Prostate Cancer
Brief Title: AMG 102 in Combination With Mitoxantrone and Prednisone in Subjects With Previously Treated Castrate Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20070611
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-02

CONDITIONS: Cancer; Castrate-Resistant Prostate Cancer; Mestastatic Prostate Cancer; Prostate Cancer
Keywords: CRPC
MeSH Terms: conditions — Neoplasms; Prostatic Neoplasms | interventions — rilotumumab; Mitoxantrone; Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Phase 1b - AMG 102 (Other): Phase 1b is an open-label study with AMG 102 at 15mg/kg de-escalating to 7.5mg/kg and 5mg/kg if needed, will be administered by IV Q3W in combination with MP.
  Interventions: Drug: AMG 102; Drug: Mitoxantrone; Drug: Prednisone
- Phase 2 Arm A - AMG 102 + MP (Experimental): AMG 102 safe dose level in phase 1b in combination with MP, will be administered by IV Q3W.
  Interventions: Drug: AMG 102; Drug: Mitoxantrone; Drug: Prednisone
- Phase 2 Arm C- PLACEBO (Placebo Comparator): Placebo in combination with MP, will be administered by IV Q3W.
  Interventions: Drug: Mitoxantrone; Drug: Placebo; Drug: Prednisone
- Phase 2 Arm B - AMG 102 + MP (Experimental): Safe dose level in phase 1b of AMG 102 + MP will be administered by Q3W
  Interventions: Drug: AMG 102; Drug: Mitoxantrone; Drug: Prednisone

INTERVENTIONS:
Drug: AMG 102 — Investigational product to be given at safe dose from phase 1b, will be administered by IV Q3W.
  Other Names: Rilotumumab
  Arms: Phase 2 Arm A - AMG 102 + MP; Phase 2 Arm B - AMG 102 + MP
Drug: AMG 102 — Investigational product to be given at 15mg/kg, 7.5mg/kg, or 5mg/kg depending on assignment, will be administered by IV Q3W.
  Other Names: Rilotumumab
  Arms: Phase 1b - AMG 102
Drug: Mitoxantrone — Administered Q3W for a maximum of 12 cyles
Drug: Placebo — Placebo
  Arms: Phase 2 Arm C- PLACEBO
Drug: Prednisone — 5 mg orally BID

SUMMARY:
The primary objectives of this study are the following:

Phase 1b: To identify a safe dose level of AMG 102, up to 15 mg/kg Q3W, to combine with mitoxantrone and prednisone (MP) Phase 2: To estimate with adequate precision the effect of the addition of AMG 102 to MP, compared with placebo plus MP, as assessed by the hazard ratio (HR) for overall survival (OS) of previously treated subjects with castrate-resistant prostate cancer (CRPC)

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed adenocarcinoma of the prostate
* Radiographic evidence of metastatic disease
* Progressive disease meeting at least one of the following criteria:

  1. a sequence of at least 2 rising PSA values measured at a minimum of 1 week apart with a 2 ng/mL minimum starting value, or
  2. progression according to RECIST criteria for measurable lesions, or
  3. appearance of 2 or more new lesions on bone scan.
* History of prior taxane-based chemotherapy for metastatic prostate cancer
* For patients without a history of surgical castration, continued GnRH analog administration is required
* ECOG Performance status of 0 or 1
* Life expectancy ≥ 3 months

Exclusion Criteria:

* Treatment with external beam radiotherapy ≤ 14 days before enrollment or radiopharmaceutical ≤8 weeks
* ≤ 4 weeks since receipt of most recent prior chemotherapy, non-GnRH analog hormonal therapy (except for continuing corticosteroids) or other systemic therapy to treat prostate cancer and <6 weeks since receipt of prior bevacizumab.
* Known CNS metastases (epidural disease is allowed if it has been treated and there is no progression in the treated area).
* Significant cardiovascular disease
* LVEF < 50% by MUGA or ECHO
* Treatment of infection with systemic anti-infectives within 7 days before enrollment (with the exception of uncomplicated urinary tract infection)
* Concurrent or prior (within 7 days of enrollment) anticoagulation therapy, except that use of low dose coumarin-type anticoagulants or heparins for prophylaxis against central venous catheter thrombosis is allowed
* Major surgical procedure ≤30 days before enrollment or not yet recovered from prior major surgery
* Presence of peripheral edema > Grade 2
* Known positive test for HIV, hepatitis C, chronic or active hepatitis B
* Serious or non-healing wound
* Unable to begin protocol specified treatment within 7 days after enrollment
* Other investigational procedures are excluded.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2008-11; Primary Completion 2011-01 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Phase 1b - Incidence of adverse events defined by dose-limiting toxicities | 21 days after the 6th subjects has recieved 1st cycle of AMG 102 in combination with MP
Phase 2 - Overall survival | Entire Study

SECONDARY OUTCOMES:
Phase 1b - Incidence of adverse events, abnormal laboratory values not defined as dose limiting toxicities | Treatment Period
Phase 1b - Incidence of anti-AMG 102 antibody formation | Entire Study
Phase 1b - Cmax and Cmin of AMG 102 concentration | Treatment Period
Phase 2 - Progression-free survival | Entire Study
Phase 2 - Maximum percentage reduction in PSA level | Entire Study
Phase 2 - PSA response rate (≥50% reduction in PSA values from baseline) | Entire Study
Phase 2 - Objective response rate (CR and PR per RECIST with modifications) | Entire Study
Phase 2 - Patient Report Outcome including pain-specific measures | Treatment Period
Phase 2 - Incidence of adverse events and significant laboratory value changes from baseline | Treatment Period
Phase 2 - Incidence of anti-AMG 102 antibody formation | Entire Study
Phase 2 - Cmax and Cmin of AMG 102; Cmax and AUC for Mitoxantrone | Treatment Period
Phase 2 - Percentage change in PSA levels from baseline to 12 weeks (or earlier for those who discontinue therapy) | Treatment Period

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Oliner K.BM Ph2 CRPC.Journal-004521;
- [Background] Ryan CJ, Rosenthal M, Ng S, Alumkal J, Picus J, Gravis G, Fizazi K, Forget F, Machiels JP, Srinivas S, Zhu M, Tang R, Oliner KS, Jiang Y, Loh E, Dubey S, Gerritsen WR. Targeted MET inhibition in castration-resistant prostate cancer: a randomized phase II study and biomarker analysis with rilotumumab plus mitoxantrone and prednisone. Clin Cancer Res. 2013 Jan 1;19(1):215-24. doi: 10.1158/1078-0432.CCR-12-2605. Epub 2012 Nov 7. PMID 23136195
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com